CLINICAL TRIAL: NCT03028883
Title: Relationship Between Buprenorphine Dose Adjustments and Gestational Age in the Treatment of Opioid-Maintained Pregnant Women
Brief Title: Buprenorphine Dose Adjustments and Gestational Age
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jaye Shyken, MD, Principal Investigator, St. Louis University
Other Study IDs: 27675
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- buprenorphine dose adjustments: To determine if a relationship exists between buprenorphine dose adjustments and gestational age in opioid-maintained pregnant women
  Interventions: Other: Dose adjustments

INTERVENTIONS:
Other: Dose adjustments — Do higher doses of buprenorphine result in a higher rate of neonatal abstinence syndrome as compared to lower doses of buprenorphine
  Other Names: buprenorphine dose adjustments

SUMMARY:
In this retrospective cohort study, we plan to examine the relationship between buprenorphine dose adjustments, gestational age, urine buprenorphine levels and the rate of neonatal abstinence syndrome in opioid-maintained pregnant women

DETAILED DESCRIPTION:
The prevalence of opioid use disorder in pregnancy was four per 1000 deliveries in 2011 and has increased to 5.4% in 2013. Repeated, acute withdrawal during pregnancy is not recommended as it is may be associated with intrauterine growth restriction (IUGR) and preterm labor and delivery. The American College of Obstetricians and Gynecologists (ACOG) recommends methadone as the first line treatments for opioid use during pregnancy and buprenorphine as an alternative. Methadone therapy has been used since the 1970's for the treatment of heroin addiction during pregnancy and efficacy is well documented. Prescribing methadone has barriers, such as significant drug interactions and enrollment in a registered substance abuse treatment program. Emerging evidence supports the use of buprenorphine for opioid use disorder in pregnancy. Buprenorphine has some distinct advantages over methadone which include a lower risk of overdose, fewer drug interactions, and no need for registration into a methadone treatment program. However, buprenorphine has a lower rate of retention in treatment than methadone.

Opioid use disorder increases the risk of adverse pregnancy outcomes compared to women who do not use opioids.One such outcome is neonatal abstinence syndrome (NAS) which affects approximately 55% to 94% of neonates exposed to addictive medications during pregnancy. A 2016 review of five trials involving buprenorphine and methadone in pregnant patients found that buprenorphine significantly improved or had similar outcomes to methadone for neonatal outcomes. Buprenorphine exposed infants required less treatment for NAS (20%-47% vs 45.5%-57%, respectively) and experienced a shorter duration of NAS (4.1-5.6 vs 5.3-9.9 days, respectively) compared to methadone exposed infants. Buprenorphine is associated with fewer preterm deliveries and adverse fetal outcomes including the rate of NAS, medication assistance for NAS, and total dose of morphine used to treat NAS. There are currently no studies evaluating the level of buprenorphine doses on the rate of NAS.

Several pharmacokinetic changes occur during pregnancy which impact medications and increase the risk for subtherapeutic levels. Subtherapeutic buprenorphine levels may increase the risk for withdrawal symptoms and cravings, which may increase the risk for relapse. The volume of distribution increases for both hydrophilic and lipophilic medications throughout pregnancy due to increased body fluid, increased adipose tissue, and decreased protein binding. Buprenorphine is metabolized through cytochrome P450 (CYP450) 3A4, UGT1A1, 1A3, and 2B7. Pregnancy increases hepatic metabolism of the CYP450 3A4 and UGT2B7. Buprenorphine is eliminated 70% through the feces and 30% through the urine. Pregnancy increases hepatic and renal elimination. Elimination is increased partly due to increased cardiac output secondary to increased plasma volume. Cardiac output reaches its maximum at approximately 32 weeks, whereas peak renal elimination occurs at 36 weeks. These pharmacokinetic changes typically require doses to be increased as pregnancy progresses.

A limitation of methadone therapy is the unpredictable pharmacokinetics during pregnancy. Methadone is a lipophilic and highly protein-bound medication, making the medication less available during pregnancy. It is metabolized mainly by CYP3A4, which leads to decreased concentrations of methadone in the plasma during pregnancy. One study performed by Pond and colleagues examined methadone serum concentrations during the second and third trimesters and at two separate time points post-partum. They found plasma trough methadone concentrations were lower and methadone renal clearance was higher in the second and third trimesters than in the post-partum time period, supporting the finding that methadone requires dose increases as pregnancy progresses. A literature review explored studies related to dosing and monitoring of methadone in pregnancy. This review included a a study that found a methadone plasma trough level of 0.78 µmol/L was required to prevent withdrawal. The authors of the review found evidence to support that methadone pharmacokinetics appear to be altered in pregnancy but that there is a lack of evidence to support routine serum monitoring. Although based on the Drozdick study they do endorse monitoring trough levels when withdrawal symptoms are apparent.

Few studies evaluated the effect of pregnancy on the pharmacokinetics of buprenorphine. Based on the characteristics of the medication it would be expected that pharmacokinetic changes in pregnancy would be similar to those of methadone. One difference is that buprenorphine has an active metabolite which may make buprenorphine dosing more predictable. the pharmacokinetics of buprenorphine in plasma, oral fluid, and sweat of pregnant women (n=9). At 28-29 and 34 weeks gestation and 2 months postpartum, plasma, oral fluid and sweat levels were collected over 24 hours. The maximum concentration and total amount of buprenorphine and norbuprenorphine in plasma were lower during pregnancy compared with postpartum levels (buprenorphine Cmax 0.2ng/mL/mg vs 1ng/mL/mg and Tmax 1.5h*ng/mL/mg vs 7h*ng/mL/mg, norbuprenorphine Cmax 3ng/mL/mg vs 13ng/mL/mg and Tmax no change). Therefore, these significant metabolic changes during pregnancy and immediately postpartum could indicate the need for dose adjustment of buprenorphine. Another small trial of nine pregnant women on buprenorphine maintenance therapy assessed the urinary excretion of buprenorphine and its metabolites every 12 days from the second trimester through 6 weeks postpartum. The mean ratio of urine buprenorphine to norbuprenorphine was significantly higher in the second trimester compared to the third trimester in all patients. Additionally, the mean dose of buprenorphine increased from the second to the third trimester in seven of the nine women. In a subset of 3 patients, 24-hour buprenorphine and metabolite excretion was collected. Buprenorphine levels were higher during pregnancy than postpartum in all three (0.8 mg, 5.0 mg, 2.0 mg vs 0.55 mg, 4.0 mg, 0.8 mg, respectively). The uncorrected buprenorphine urine concentrations ranged from 5.5 to 12.1 µg/L [mean 7.0 (2.8) µg/L], although they did not evaluate if withdrawal symptoms occurred below a certain threshold. The buprenorphine dose in this study was flexible, with increases or decreases made through clinical decisions based on compliance in taking medication, participant requests, urine toxicology, and participant self-reports of opioid withdrawal symptoms or craving. Buprenorphine dose was positively correlated to creatinine-corrected norbuprenorphine (P < 0.001, R = 0.197), buprenorphine-glucuronide (P < 0.002, R = 0.143), and norbuprenorphine-glucuronide (P < 0.001, R = 0.182) concentrations across the study. However low correlation coefficients indicate that prediction of metabolite concentrations in urine based on buprenorphine dose, or vice versa, would be unreliable. These studies support the need for increased doses of buprenorphine throughout pregnancy, but may have been too small to determine whether a relationship between buprenorphine urine levels and dose adjustments exists. Currently, no studies examined the relationship between gestational age and buprenorphine dose adjustments after having achieved maintenance dosing.

This information could assist providers in optimizing monitoring of pregnant women and informing providers regarding dose adjustments. Preventing subtherapeutic levels may decrease the risk for withdrawal symptoms, craving, and risk of relapse.

No data are available to evaluate whether a particular gestational age requires dose adjustments due to pregnancy-related pharmacokinetic changes. The program obtains quantitative and qualitative buprenorphine and norbuprenorphine urine levels at each visit. These data are used to confirm that she is taking her buprenorphine prescription. No data are available to determine if there is a lower threshold in urine buprenorphine and metabolite that levels correlate with symptoms that require dose increases. Additionally, no data are available evaluating if rates of NAS, treatment for NAS, or total dose of morphine for NAS correlates as a function of maternal dose.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* opioid-dependent
* being treated at same location

Exclusion Criteria:

* Not pregnant
* not opioid-dependent

Ages: 14 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ages 14-55yrs of age Female any ethnic background
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
dose adjustments | 9 months
  buprenorphine dose adjustments in opioid-maintained pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Jaye Shyken, MD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No